CLINICAL TRIAL: NCT02093832
Title: Does the Femoral Head Size Can Predict the Cup Size? Retrospective Study.
Brief Title: Does the Femoral Head Size Can Predict the Cup Size?
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 0067-13-EMC
Record Dates: First submitted 2014-03-11; First posted 2014-03-21 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Total Hip Arthroplasty
Keywords: femoral head size; cup size; Total hip arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Total hip arthroplasty
  Interventions: Other: There are no specific Intervention

INTERVENTIONS:
Other: There are no specific Intervention — are no specific Intervention
  Other Names: are no specific Intervention

SUMMARY:
This study had four aims:

1. To evaluate the correlation between the planned preoperative cup size and the actual cup size that was implanted in surgery.
2. To examine the absolute difference between the implanted cup size diameter and the actual femoral head size diameter.
3. To examine the absolute difference between the planned cup size diameter and the actual femoral head size diameter
4. To suggest an additional online monitoring tool on the accuracy of the preoperative process and implant selection. We hypothesized that high accuracy rates will be found between the preoperative planned cup size and the actual implanted cup size. Furthermore, we hypothesized that strong correlations will be found between the planned and actual implanted cup size and the actual femoral head diameter size.

DETAILED DESCRIPTION:
Methods This is a retrospective study , that will include patients who underwent primary cementless THA due to end-stage hip osteoarthritis during 2011 and 2013 . Inclusion criteria were: Patients that underwent primary THA due to end-stage primary osteoarthritis; Males and females between 15-90 years of age.

Data collection The following data will be collected: patients' characteristic including gender, age at surgery and side of surgery; implant information including cup model, planed cup size, actual cup size, shell type and outer diameter size (mm); actual femoral head diameter size (mm); the difference between the planned cup size and the actual cup size that was used; the difference between the actual femoral head diameter size measured at the end of surgery and the cementless implanted cup outer diameter size; the difference between the actual femoral head diameter size and the planed cup size..

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent primary Total hip arthroplasty due to end-stage primary osteoarthritis;

Exclusion Criteria:

* Significant distortion in the femoral head.
* Previous reconstructive surgery - radial osteotomy and hip socket.

Ages: 15 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent primary Total hip arthroplasty due to end-stage primary osteoarthritis; Males and females between 15-90 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the correlation between the planned preoperative cup size and the actual cup size that was implanted in surgery. | up to one year

SECONDARY OUTCOMES:
To examine the absolute difference between the implanted cup size diameter and the actual femoral head size diameter. | up to one year

OTHER OUTCOMES:
To examine the absolute difference between the planned cup size diameter and the actual femoral head size diameter | up to one year

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - HeEmek medical center, Afula
  - Orthopedic department, HaEmek medical center, Afula